CLINICAL TRIAL: NCT00929227
Title: Comparison of Cardiac Computed Tomography and Vasodilator Stress Magnetic Resonance Imaging Perfusion in Patients With Prior Equivocal Stress Test for Detection of Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090164; 09-H-0164
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Coronary Artery Disease
Keywords: Inconclusive Noninvasive Cardiac Stress Test; Cardiac Computed Tomography; Coronary Artery Disease; Atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Stress MRI perfusion, and cardiac CT will have observed sensitivity, specificity, and accuracyof at least 0.80 in predicting CAD in a patient population with prior equivocal stress testing.

SUMMARY:
Background:

* Noninvasive cardiac stress testing is imperfect. Inconclusive test results generate further expensive testing.
* In patients with known or suspected coronary artery disease, both computed tomography (CT) and magnetic resonance imaging (MRI) have been shown to provide suitable results for detecting the disease. However, both types of scans have limitations in their usefulness, and it is not known whether one is preferable in either accuracy or cost-effectiveness.

Objectives:

- To determine the accuracy and cost-effectiveness of CT and MRI in subjects with a prior inconclusive heart stress test.

Eligibility:

- Patients 18 years of age and older who have had an inconclusive heart stress test within the past 90 days.

Design:

* A blood test will be obtained prior to both heart tests. This will require less than a teaspoon of blood.
* A CT scan will be performed, accompanied by beta blocker medications (to slow heart rate) or nitroglycerin (to enlarge blood vessels) to improve picture quality, as needed.
* An MRI scan will be performed. Scans will be taken before, during, and after the patient receives vasodilators (to increase blood flow to the coronary arteries and detect blockages in heart blood vessels).
* Heart rate and function will be monitored with an electrocardiogram.

DETAILED DESCRIPTION:
Noninvasive cardiac stress testing is imperfect. Inconclusive test results generate further expensive testing. We will do both cardiac computed tomography (CT) and stress cardiac magnetic resonance imaging (MRI) in patients who have an inconclusive noninvasive cardiac stress test. We will test whether MRI predicts significant coronary artery disease in a more cost-effective and accurate manner than CT, or vice versa.

ELIGIBILITY:
* GENERAL INCLUSION CRITERIA:
* 18 years of age and older
* Prior equivocal stress study within the preceding 90 days
* Able to provide informed consent

MEDICAL EXCLUSION CRITERIA:

* Decompensated heart failure (unable to lie flat during MRI or CT)
* Severe kidney disease (MDRD estimated Glomerular Filtration Rate less than 30mL/min/1.73m(2).
* Prior cardiac revascularization with coronary stent or bypass surgery
* Resting tachycardia (HR greater than l00 bpm)
* Pregnant women (when uncertain, subjects will undergo urine or blood testing)
* Lactating women (unless they are willing to discard breast milk for 24 hours after receiving gadolinium)
* Second (Type II) and third degree atrioventricular heart block
* Asthma or chronic pulmonary disease (emphysema) actively treated with bronchodilators or leukotriene antagonists

MRI EXCLUSION CRITERIA:

* Cardiac pacemaker or implantable defibrillator
* Cerebral aneurysm clip
* Neural stimulator (e.g. TENS-Unit)
* Any type of ear implant
* Ocular foreign body (e.g. metal shavings)
* Any implanted device (e.g. insulin pump, drug infusion device)
* Metal shrapnel or bullet

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This trial will involve the NIH Clinical Center and Suburban Hospital. Subjects with an equivocal stress study determined by a referring physician will be recruited from the surrounding community.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2020-11-19 (Actual)

PRIMARY OUTCOMES:
Stress MRI perfusion, and cardiac CT will have observed sensitivity, specificity, and accuracy of at least 0.80 in predicting CAD in a patient population with prior equivocal stress testing. | end of study
  estimate the sensitivity, specificity, and accuracy of MRI and CT, for detecting obstructive CAD in patients with a prior equivocal stress study

SECONDARY OUTCOMES:
The null hypothesis is that there will be no difference between stress MRI perfusion and cardiac CT with respect to the diagnostic costs for patients with an equivocal stress study for CAD. | end of study
  compare the cost-effectiveness of MRI with CT for this patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Sirajuddin, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (2):
- United States (2):
  - Suburban Hospital, Bethesda, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Hendel RC, Wackers FJ, Berman DS, Ficaro E, DePuey EG, Klein L, Cerqueira M; American Society of Nuclear Cardiology. American Society of Nuclear Cardiology consensus statement: Reporting of radionuclide myocardial perfusion imaging studies. J Nucl Cardiol. 2006 Nov;13(6):e152-6. doi: 10.1016/j.nuclcard.2006.08.013. No abstract available. PMID 17174791
- [Background] Brindis RG, Douglas PS, Hendel RC, Peterson ED, Wolk MJ, Allen JM, Patel MR, Raskin IE, Hendel RC, Bateman TM, Cerqueira MD, Gibbons RJ, Gillam LD, Gillespie JA, Hendel RC, Iskandrian AE, Jerome SD, Krumholz HM, Messer JV, Spertus JA, Stowers SA; American College of Cardiology Foundation Quality Strategic Directions Committee Appropriateness Criteria Working Group; American Society of Nuclear Cardiology; American Heart Association. ACCF/ASNC appropriateness criteria for single-photon emission computed tomography myocardial perfusion imaging (SPECT MPI): a report of the American College of Cardiology Foundation Quality Strategic Directions Committee Appropriateness Criteria Working Group and the American Society of Nuclear Cardiology endorsed by the American Heart Association. J Am Coll Cardiol. 2005 Oct 18;46(8):1587-605. doi: 10.1016/j.jacc.2005.08.029. PMID 16226194
- [Background] Hendel RC, Patel MR, Kramer CM, Poon M, Hendel RC, Carr JC, Gerstad NA, Gillam LD, Hodgson JM, Kim RJ, Kramer CM, Lesser JR, Martin ET, Messer JV, Redberg RF, Rubin GD, Rumsfeld JS, Taylor AJ, Weigold WG, Woodard PK, Brindis RG, Hendel RC, Douglas PS, Peterson ED, Wolk MJ, Allen JM, Patel MR; American College of Cardiology Foundation Quality Strategic Directions Committee Appropriateness Criteria Working Group; American College of Radiology; Society of Cardiovascular Computed Tomography; Society for Cardiovascular Magnetic Resonance; American Society of Nuclear Cardiology; North American Society for Cardiac Imaging; Society for Cardiovascular Angiography and Interventions; Society of Interventional Radiology. ACCF/ACR/SCCT/SCMR/ASNC/NASCI/SCAI/SIR 2006 appropriateness criteria for cardiac computed tomography and cardiac magnetic resonance imaging: a report of the American College of Cardiology Foundation Quality Strategic Directions Committee Appropriateness Criteria Working Group, American College of Radiology, Society of Cardiovascular Computed Tomography, Society for Cardiovascular Magnetic Resonance, American Society of Nuclear Cardiology, North American Society for Cardiac Imaging, Society for Cardiovascular Angiography and Interventions, and Society of Interventional Radiology. J Am Coll Cardiol. 2006 Oct 3;48(7):1475-97. doi: 10.1016/j.jacc.2006.07.003. No abstract available. PMID 17010819
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-H-0164.html